CLINICAL TRIAL: NCT05800639
Title: Mediation Role of Perioperative Electroencephalogram Frontal Alpha Asymmetry to Pediatric Emergence Delirium
Brief Title: Frontal Alpha Asymmetry and Pediatric Emergence Delirium
Status: Recruiting | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Young Song, Professor, Gangnam Severance Hospital
Other Study IDs: 3-2023-0014
Record Dates: First submitted 2023-03-24; First posted 2023-04-05 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Emergence Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Ophthalmologic Surgical Procedures; Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with emergence delirium: Pediatric patients who develop emergence delirium in the post-anesthetic care unit (PACU).
  Emergence delirium will be assessed using the Pediatric Assessment of Emergence Delirium (PAED) scale every 10 min until PACU discharge.
  Interventions: Procedure: Ophthalmic surgery; Procedure: General anesthesia
- Children without emergence delirium: Pediatric patients who do not develop emergence delirium in the post-anesthetic care unit (PACU).
  Emergence delirium will be assessed using the Pediatric Assessment of Emergence Delirium (PAED) scale every 10 min until PACU discharge.
  Interventions: Procedure: Ophthalmic surgery; Procedure: General anesthesia

INTERVENTIONS:
Procedure: Ophthalmic surgery — Ophthalmic surgery will be performed as standard practice of our institution.
Procedure: General anesthesia — General anesthesia will be performed as standard practice of our institution.

SUMMARY:
This study aimed to investigate whether the association between the preoperative anxiety level and emergence delirium involves EEG frontal alpha asymmetry in pediatric patients undergoing ophthalmic surgery under general anesthesia. The investigators hypothesized that EEG frontal alpha asymmetry contributes a significant portion of the preoperative anxiety - emergence delirium association in pediatric patients. Mediation analysis will be performed to estimate the relationships between preoperative anxiety of children (modified Yale Preoperative Anxiety Scale (mYPAS)), EEG frontal alpha asymmetry, and emergence delirium (Pediatric Assessment of Emergence Delirium (PAED) scale).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2-8 year
* Children with an American Society of Anesthesiologists (ASA) physical status of I-II
* Children who are scheduled to undergo elective ophthalmological requiring general anesthesia

Exclusion Criteria:

* Emergency surgery
* Patients with developmental delays
* Patients with neurological or psychiatric diseases associated with symptoms of agitation, anxiety, attention deficit, sleep disturbances
* Patients with autism
* Patients with a recent history (within one month) of receiving general anesthesia
* Patients with congenital or genetic diseases that may influence brain development

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 2-8 year with an American Society of Anesthesiologists (ASA) physical status of I-II who are undergoing elective ophthalmological requiring general anesthesia in Gangnam Severance Hospital will be eligible.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
The peak PAED score | After the completion of surgery, during the PACU stay. PAED score will be measured every 10 minutes during the PACU stay.
  The peak PAED score is the primary outcome variable for mediation analysis

CONTACTS AND LOCATIONS:
Overall Officials: Young Song, Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea